CLINICAL TRIAL: NCT02242292
Title: A Double-blind, Placebo-controlled, Randomized, Parallel Group Study of the Efficacy and Safety of Oral Doses of 20 mg Hyoscine Butylbromide When Used On-demand up to 7 Episodes Over a Period of 6 Weeks for the Treatment of Occasional Episodes of Self-reported Abdominal Pain, Cramping, and Discomfort Associated With Cramping in an OTC-like Study Population
Brief Title: Study to Evaluate Efficacy and Safety of Oral Doses of Hyoscine Butylbromide for the Treatment of Occasional Abdominal Pain, Cramping, and Discomfort
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202.832
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Colic
MeSH Terms: conditions — Colic | interventions — Butylscopolammonium Bromide

ARMS (2):
- Hyoscine butylbromide (Experimental): 5 tablets taken in a 24-hour period/each episode:
  * for up to 7 episodes, or
  * over a period of up to 6 weeks
  Interventions: Drug: Hyoscine butylbromide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hyoscine butylbromide
  Arms: Hyoscine butylbromide
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to determine whether hyoscine butylbromide can provide adequate symptomatic relief of a single episode - defined as lasting not longer than 1 day - and multiple episodes of abdominal pain or discomfort associated with cramping when used as needed

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females 18 years of age and older
2. Have at least a 3-month self-reported history of recurrent episodic symptoms, usually lasting for 1 hour or more, of self-described abdominal pain or discomfort associated with cramping, which they routinely either have not treated or treated using Over-the-counter (OTC) medications, in which subjects suffered these symptoms at a frequency of at least twice monthly to several times weekly, but not on a daily basis. The episodes of abdominal pain or discomfort may have been associated with other symptoms of GI dysfunction, such as diarrhea, constipation, and bloating
3. Symptoms typically have a moderate or greater severity (moderate, severe, very severe) and are sufficiently bothersome to require treatment or intervention
4. Symptoms are not associated with abdominal tenderness, swelling, fever, weight loss, or passage of blood per rectum. The onset of symptoms may or may not have been associated with ingestion of food or beverages
5. The episodes of abdominal pain or discomfort may have been associated with other symptoms of GI dysfunction, such as diarrhea, cramping, constipation, and bloating
6. Subjects are required to be able to comprehend and participate in the activities required for participation in the trial, to have the ability to attend required site visits, and to be available and have the facility to participate in a daily telephone call or computer entry (using a touch-tone phone or computer IVRS entry), which served as the mechanism for diary entry, during the 6-week course of the study. Subjects were required to successfully complete an Interactive voice response system (IVRS) training session prior to entry into the study
7. All subjects completed and signed an informed consent form

Exclusion Criteria:

1. Subjects who reported having these symptoms for the first time, particularly if they were 50 years or older, as this may have been a sign of a more serious organic disease
2. Subjects with a known hypersensitivity or allergy to hyoscine butylbromide or any of the inactive ingredients
3. Subjects who are currently under a physician's care for abdominal symptoms and/or not using medication or using prescription or OTC medications prescribed by a physician to treat symptoms of abdominal pain, cramping and discomfort or taking prescription medication(s) for the treatment of Irritable bowel syndrome (IBS) (Bentyl® or other antispasmodics, Zelnorm® [tegaserod], Lotronex® [alosetron], prokinetic agents). Current physician's care was defined as the subject presently following clinician advice regarding treatment and management of the abdominal pain or discomfort associated with the cramping symptom
4. Subjects who are having symptoms of abdominal swelling, fever associated with symptoms of abdominal pain or discomfort associated with cramping, and/or experiencing passage of blood per rectum associated with symptoms of abdominal pain or discomfort associated with cramping, or who have any evidence of abdominal tenderness (or any other evidence of an acute abdomen), abdominal masses, organomegaly or any other abnormality on abdominal examination
5. Subjects with a history of colon or other GI cancer or malignancy, inflammatory bowel disease, or Crohn's disease
6. Subjects with chronic constipation
7. Subjects with myasthenia gravis or megacolon
8. Subjects who have undergone abdominal surgery within the past 2 years, having GI surgery resulting in removal of all or part of the colon, small intestine, or stomach, or having a history of GI by-pass surgery for weight reduction
9. Prior history of gallbladder removal, appendectomy, and/or surgery for peptic ulcer disease or gastroesophageal reflux disease (GERD), was not exclusionary.
10. Subjects whose major symptoms were retrosternal burning, acid reflux, acid regurgitation, or heartburn are excluded
11. Subjects using prescription anticholinergic medications or medications for the treatment of myasthenia gravis, glaucoma, or ocular hypertension are excluded
12. Subjects who were currently participating in other trials or who participated in a clinical trial within the prior 30 days are excluded
13. Women who reported being pregnant, are nursing, or who are of child-bearing potential and not using an adequate method of birth control (medication, device, abstinence, sterilization for either partner) for 30 days before enrollment and did not agree to continue using an adequate method of birth control for 30 days after completion of the trial are excluded
14. Any women of childbearing potential who have a positive serum pregnancy test are excluded
15. Post-menopausal women who have been post-menopausal for a duration of less than 2 years and did not have a hysterectomy or tubal ligation procedure are excluded
16. Subjects who have tachyarrhythmia (defined as any disturbance of the heart's rhythm, regular or irregular, resulting in a rate over 100 beats per minute) during a physical examination are excluded
17. Subjects who have been previously diagnosed with benign prostatic hyperplasia (BPH) or subjects who experienced urinary retention are excluded
18. Subjects with clinically significant cardiovascular disease in the opinion of the investigator (including hypotension, hypertension, severe coronary artery disease, congestive heart failure, angina pectoris) are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2006-04; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Response rate in treating the first episode of abdominal pain or discomfort associated with cramping | within 24 hours after starting treatment
  (Response was defined as achieving adequate relief of symptoms, as measured on a subject's diary using a dichotomized response to the question)

SECONDARY OUTCOMES:
Response rate to trial medication | up to day 41
  responders were those who obtained adequate relief for 50% or more of all treated episodes
Assessment of Average symptom relief rated on 4-point scale | up to day 41
  based on the "Symptom Relief Index''
Time to onset of any effect after the first tablet taken assessed on 5-point scale | within 24 hours after starting treatment
Time to onset of any effect assessed on 5-point scale | up to day 41
Time to obtain adequate relief after the first tablet taken assessed on 5-point scale | within 24 hours after starting treatment
Time to obtain adequate relief assessed on 5-point scale | up to day 41
Average time to obtain adequate relief per subject assessed on 5-point scale | up to day 41
Average number of tablets taken to treat episodes per subject | up to day 41
  measured for each treated episode by the subject's response to the question on the number of tablets taken for each treated episode or 24-hour period
Percentage of episodes of diarrhea | up to day 41
Percentage of bloating episodes | up to day 41
Percentage of constipation episodes | up to day 41
Percentage of episodes in relief of abdominal pain or discomfort associated with cramping | up to day 41
Global Assessment of efficacy by subject on 4-point scale | Day 42
Global Assessment of tolerability by subject on a 4-point scale | Day 42
Global assessment of tolerability by investigator on a 4- point scale | Day 42
Number of patients with adverse events | up to 42 days
Number of patients with abnormal changes in laboratory parameters | up to 42 days

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/16817918